CLINICAL TRIAL: NCT00057694
Title: Genetic Information: Exploring the Value to Adult Adoptees
Brief Title: The Value of Genetic Information to Adult Adopted Individuals
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030144; 03-HG-0144
Record Dates: First submitted 2003-04-05; First posted 2003-04-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-01

CONDITIONS: Adoption; Genetic Counseling
Keywords: Qualitative; Telephone Interviews; Genetic Counseling; Family History; Health Information; Adult Adoptees; Adult Adoptee; Interview

SUMMARY:
This study will explore adult adoptees' perceptions of the potential value of genetic and family history information. Unlike most people, many adopted individuals do not have access to personal or family medical information because of laws and practices that prevent disclosure. Research suggests that adopted individuals are interested in obtaining this information about their biological families. This study will examine adoptees':

* Satisfaction with the amount of genetic information they have, their motivations for wanting more information, and when it becomes important for them to have this information.
* Perceptions of the degree to which they believe genetics and family history influence various traits and conditions.

The study will also explore adoptees' interactions with health care providers so that recommendations can be developed for helping genetic counselors meet the needs of these individuals.

English-speaking adoptees 18 years of age and older are eligible for this study. Those enrolled will participate in a one-time telephone interview that will take about 45 to 60 minutes. The interview will obtain demographic information, such as the adoptee's age, sex, racial and ethnic background, marital status, and education level, and will include questions in the following areas:

* Personal adoption story;
* Perceptions of the role of the biological family history and medical information and its importance and usefulness;
* Perceptions of the influence of genetics and family history on health;
* Reproductive history and pregnancy concerns related to being adopted;
* Experiences and interactions with health care providers related to adoption;
* Suggestions for improving interactions with health care providers.

DETAILED DESCRIPTION:
In contrast to the majority of the population, many adopted individuals do not have access to personal or familial medical information because of laws and practices that prevent disclosure. A body of research has suggested however that adopted individuals are interested in obtaining this information regarding their biological families. The proposed study broadly aims to explore adult adoptees' perceptions regarding the potential value of genetic and family history information. Specifically it will investigate adoptees' motivations for obtaining the information, their perceptions regarding the influence of genetics on health, and their experiences with healthcare providers related to adoption and medical information. These objectives will be addressed in telephone interviews with English-Speaking adult adoptees (over the age of 18 years) that were placed in unrelated adoptive families. A semi-structured guide for the telephone interviews consists of a series of open-ended questions that explore the objectives of the study. We hope to collect data on about 40 individuals. The data will be subject to coding for thematic analyses to identify recurring trends and themes. This study has implications for genetic counselors as the findings may guide the development of appropriate educational messages and counseling recommendations for adopted individuals related to their genetic and family history information.

ELIGIBILITY:
INCLUSION CRITERIA:

English-speaking adoptees, over 18 years of age, who were placed in unrelated adoptive families.

EXCLUSION CRITERIA:

Adult adoptee that participated in piloting.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-04; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States

REFERENCES:
- [Background] American Society of Human Genetics Social Issues Committee report on genetics and adoption: points to consider. Am J Hum Genet. 1991 May;48(5):1009-10. No abstract available. PMID 2018032
- [Background] Aumend SA, Barrett MC. Self-concept and attitudes toward adoption: a comparison of searching and nonsearching adult adoptees. Child Welfare. 1984 May-Jun;63(3):251-9. PMID 6723422
- [Background] Bansal A, Critchfield GC, Frank TS, Reid JE, Thomas A, Deffenbaugh AM, Neuhausen SL. The predictive value of BRCA1 and BRCA2 mutation testing. Genet Test. 2000;4(1):45-8. doi: 10.1089/109065700316462. PMID 10794360